CLINICAL TRIAL: NCT04761601
Title: A Phase 1, First in Human, Dose-Escalation Study of UCT-01-097 in Participants With Advanced Solid Tumors
Brief Title: First in Human Study of UCT-01-097 in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Stopped for strategic business reasons. The decision to stop the study was not connected to any safety concerns, or new risk associated with the study product, intervention, or procedures.
Sponsor: 1200 Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UCT01097-001
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Gemcitabine; Paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Finding as Monotherapy - Part 1 (Experimental)
  Interventions: Drug: UCT-01-097
- Expansion as Monotherapy - Part 2 (Experimental)
  Interventions: Drug: UCT-01-097
- Dose Finding in Combination - Part 3 (Experimental)
  Interventions: Drug: UCT-01-097; Drug: Gemcitabine; Drug: Paclitaxel

INTERVENTIONS:
Drug: UCT-01-097 — Orally available kinase inhibitor
Drug: Gemcitabine — Gemcitabine injection for intravenous use.
  Other Names: Gemzar
  Arms: Dose Finding in Combination - Part 3
Drug: Paclitaxel — Paclitaxel protein-bound particles for injectable suspension (albumin-bound).
  Other Names: Abraxane
  Arms: Dose Finding in Combination - Part 3

SUMMARY:
This first-in-human study will evaluate the safety, tolerability, pharmacokinetics, and antitumor activity of UCT-01-097 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumor
* Measurable disease, per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate organ function

Exclusion Criteria:

* Has not recovered [recovery is defined as NCI CTCAE, version 5.0, grade ≤1] from the acute toxicities of previous therapy, except treatment-related alopecia or laboratory abnormalities otherwise meeting eligibility requirements
* Received prior chemotherapeutic, investigational, or other therapies for the treatment of cancer within 14 days with small molecule and within 28 days with biologic before the first dose of UCT-01-097
* Progressive or symptomatic brain metastases
* Serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection
* History of phosphate or calcium disorder
* History of significant cardiac disease
* History or current evidence/risk of retinopathy
* History of myelodysplastic syndrome (MDS) or AML
* History of another cancer within 3 years before Day 1 of study treatment, with the exception of basal or squamous cell carcinoma of the skin that has been definitively treated. A history of other malignancies with a low risk of recurrence, including appropriately treated ductal carcinoma in situ (DCIS) of the breast and prostate cancer with a Gleason score less than or equal to 6, are also not excluded
* If female, is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events and serious adverse events | up to 2 years
  Incidence and severity of adverse events, serious adverse events, according to NCI-CTCAE Version 5.0
Maximum Tolerated Dose (MTD) | 28 Days
  Highest administered dose with < 33% participants experiencing dose limiting toxicity (DLT) in the first 6 DLT evaluable participants
Recommended Phase 2 Dose (RP2D) | up to 2 years
  Based on the maximum tolerated dose, cumulative safety, and pharmacokinetic data

SECONDARY OUTCOMES:
Maximum Plasma UCT-01-097 Concentration (Cmax) | Day 1
  PK assessment for UCT-01-097
Maximum Plasma UCT-01-097 Concentration at steady state (Cmax,ss) | Day 15
  PK assessment for UCT-01-097
UCT-01-097 Trough Plasma Concentration (Cmin) | Day 1
  PK assessment for UCT-01-097
UCT-01-097 Trough Plasma Concentration at Steady State (Cmin,ss) | Day 15
  PK assessment for UCT-01-097
Time of Maximum Plasma UCT-01-097 Concentration (Tmax) | Cycle 1 (each cycle is 28 days)
  PK assessment for UCT-01-097
Area Under the Plasma Concentration-Time Curve Over Dosing Interval (AUCtau) of UCT-01-097 | Day 15
  PK assessment for UCT-01-097
Apparent Clearance (CL/F) of UCT-01-097 | Cycle 1 (each cycle is 28 days)
  PK assessment for UCT-01-097
Apparent Volume of Distribution (Vz/F) of UCT-01-097 | Cycle 1 (each cycle is 28 days)
  PK assessment for UCT-01-097
Accumulation Ratio (Rac) of UCT-01-097 | Cycle 1 (each cycle is 28 days)
  PK assessment for UCT-01-097
Terminal Half-life (t1/2) of UCT-01-097 | Cycle 1 (each cycle is 28 days)
  PK assessment for UCT-01-097
Objective Response Rate (ORR) | up to 2 years
  Percentage of participants with best response of CR or PR according to RECIST 1.1
Time to Response (TTR) | up to 2 years
  Time from start of treatment to complete response or partial response
Duration of Response (DOR) | up to 2 years
  Time from complete response or partial response to objective disease progression or death due to any cause
Progression Free Survival (PFS) | up to 2 years
  PFS is defined as the time from the start of the treatment until objective disease progression or death from any cause
1 Year Overall Survival (1YOS) | 1 year
  Proportion of participants alive at 1 year from the start of treatment to death from any cause
2 Year Overall Survival (2YOS) | 2 years
  Proportion of participants alive at 2 years from the start of treatment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Letrent, PharmD, PhD, Study Director — 1200 Pharma, LLC
Locations (6):
- United States (6):
  - UCLA - JCCC Clinical Research Unit, Los Angeles, California
  - Torrance Memorial, Torrance, California
  - Winship Institute of Emory University, Atlanta, Georgia
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Sarah Cannon, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No